CLINICAL TRIAL: NCT00012506
Title: The Safety and Efficacy of a Tumor Necrosis Factor Receptor Fusion Protein on Uveitis Associated With Juvenile Rheumatoid Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Purpose: Treatment
Other Study IDs: NEI-82
Record Dates: First submitted 2001-03-10; First posted 2001-03-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: Uveitis; Arthritis, Juvenile Rheumatoid
MeSH Terms: conditions — Uveitis; Arthritis, Juvenile | interventions — Etanercept

INTERVENTIONS:
Drug: TNFR:Fc

SUMMARY:
This study will investigate the safety and effectiveness of the drug Enbrel (TNFR:Fc) to treat uveitis (eye inflammation) in patients with juvenile rheumatoid arthritis.

DETAILED DESCRIPTION:
In other studies, TNFR:Fc significantly reduced joint pain and swelling in adult patients with rheumatoid arthritis, and the Food and Drug Administration has approved the drug for that use. Because medicines for arthritis often help patients with eye inflammation, this study will examine whether TNFR:Fc can help patients with uveitis.

Patients with uveitis who are not responding well to standard treatment, such as steroids, and patients who have side effects from other medicines used to treat their uveitis or have refused treatment because of possible side effects may be eligible for this study. Candidates will be screened with a medical history, physical examination, and eye examination. The eye exam includes a check of vision and eye pressure, examination of the back of the eye (retina), and front of the eye, including measurements of protein and inflammation. Candidates will also undergo fluorescein angiography-a procedure in which photographs are taken of the retina to see if there is any leakage in the eye's blood vessels. A blood test and joint evaluation will also be done.

Study participants will be given an injection of TNFR:Fc twice a week for up to 12 months and may continue other medicines they may be taking, such as prednisone or methotrexate. They will have follow-up examinations at week two and months one, two, three and four. Those who wish to continue treatment after the fourth month can receive the drug for another eight months and will have follow-up exams at months six, nine and 12, and one month after treatment ends. Each follow-up visit will include a repeat of the screening exams and an evaluation of side effects or discomfort from the medicine.

ELIGIBILITY:
Must meet American College of Rheumatology Criteria for JRA.

Must have active anterior uveitis defined as the presence of inflammatory cells (Grade 1+ or higher) in the anterior chamber of at least one eye or the current use of topical corticosteroids to control exacerbation of disease at a frequency of TID or higher.

Age between 2 and 18 years, inclusive.

Ability to undergo slit lamp biomicroscopy for assessment of anterior chamber cells.

Ability to comply with study requirements.

Be up to date on all recommended childhood immunizations.

Using current arthritis regimen for at least 8 weeks prior to enrollment.

No media opacity that precludes assessment of anterior chamber inflammation.

No periocular injection of corticosteroids within 2 months of baseline, or used a systemic experimental therapy within one month of baseline evaluation.

Not currently receiving disease modifying antirheumatic therapy (DMARD), with the exception of prednisone at a dose no greater than 1.0 mg/kg/day, or methotrexate at a dose no greater than 15 mg/m(2)/week.

No active eye or joint inflammation requiring immediate addition or increase in systemic anti-inflammatory medications.

No females who are pregnant or lactating.

No refusal to use contraception during the study and 6 months after termination of active study therapy, if child-bearing or fathering potential exists.

No use of Latanoprost within two weeks prior to enrollment, or have a current or likely need for Latanoprost during the course of the study.

No hypersensitivity to fluorescein dye.

No active serious infections or history of recurring serious infections.

No evidence of spondyloarthropathy or entheseopathy.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health, Bethesda, Maryland, United States